CLINICAL TRIAL: NCT01396733
Title: Clinical Trial to Evaluate Efficacy of Redifferentiation Therapy Using Alpha-lipoic Acid in Thyroid Cancer Patients With Decreased Radioactive Iodine Uptake
Brief Title: Redifferentiation Therapy Using Alpha Lipoic Acid in Thyroid Cancer
Acronym: RALT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Won Bae Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_THY_001
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Thyroid; Cancer
Keywords: thyroid; cancer; redifferentiation; lipoic acid
MeSH Terms: conditions — Thyroid Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose group (Active Comparator): Patients who will receive 600 mg/day alpha-lipoic acid
  Interventions: Drug: alpha-lipoic acids
- High dose group (Active Comparator): Patients who will receive 1,200 mg/day alpha-lipoic acid
  Interventions: Drug: alpha-lipoic acids

INTERVENTIONS:
Drug: alpha-lipoic acids — alpha-lipoic acid 600 mg/day or 1,200 mg/day 600 mg/day - Three tablets (200mg x 3), one time per day for 3 months 1,200 mg/day - Three tablets (200mg x 3), two times per day for 3 months

SUMMARY:
Radioiodine (I-131) therapy is of proven efficacy for treatment of differentiated thyroid carcinoma (DTC). However, loss of differentiation in recurrent or metastatic DTC which decrease I-131 uptake may decrease the efficacy of I-131 therapy. Therefore, strategies to improve I-131 uptake are mandatory. This study is an open label clinical study to evaluate the effectiveness of alpha-lipoic acid (ALA) for improving I-131 uptake in recurrent or metastatic of DTC with defective I-131 uptake.

ELIGIBILITY:
Inclusion Criteria:

1. aged 20 to 75 years
2. under birth control, if fertile women
3. Groups

   * who received radioactive iodine treatment for recurrent and metastatic thyroid cancer, and did not showed any uptake at post-therapeutic whole body scan
   * who planned to receive empirical radioactive treatment due to high expected recurrence

Exclusion Criteria:

* allergic to alpha-lipoic acid
* severe heart failure, lung disease, or end-stage renal disease
* liver function abnormalities (x2.5 above normal limits)
* neuropsychologically unstable patients
* previous history of drug medication such as oral steroid, digoxin, theophylline, carbamazepine, valproic acid, phenobarbital, methotrexate, cyclosporin, tacrolimus within 3 months before this recruitment.
* who is already taking alpha-lipoic acid for other purpose.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Increment of radioactive iodine uptake | 3months after alpha-lipoic acid treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea